CLINICAL TRIAL: NCT03843788
Title: Transcutaneous Electrical Nerve Stimulation and Maternal Opioid Use After Cesarean Delivery
Brief Title: TENS and Opioid Use After Cesarean Delivery
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: COVID-19 pandemic
Sponsor: Rutgers, The State University of New Jersey (Other)
Responsible Party: Principal Investigator, Adrienne Simonds PT PhD, Assistant Professor of Rehabilitation and Movement Sciences,, Rutgers, The State University of New Jersey
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Pro2018001008
Record Dates: First submitted 2018-08-07; First posted 2019-02-18 (Actual); Results first posted 2024-10-29 (Actual); Last update posted 2024-10-29 (Actual); Status verified 2024-10

CONDITIONS: Cesarean Section Complications; Opioid Use
Keywords: Post-cesarean pain; Transcutaneous Electrical Nerve Stimulation
MeSH Terms: interventions — Transcutaneous Electric Nerve Stimulation

STUDY DESIGN:
Intervention Model Description: This is a pilot feasibility study to evaluate effectiveness and acceptability in our patient population of TENS use throughout delivery hospitalization. We aim to have 20 participants total: 5 in control and 5 in intervention without history of opioid addiction, and 5 in control and 5 in intervention with history of opioid addiction/misuse. This sample size is comparable to other shorter term pilot studies. This pilot study will serve as the basis for larger trials in the future, with larger sample size powered to demonstrate reduction in pain scores. We anticipate recruitment for this trial will take approximately 6-9 months.
Masking Description: Not able to be masked
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (4):
- Post-CS TENS (Experimental): The patients in the intervention group will be educated on the proper way to utilize the transcutaneous electrical nerve stimulation (TENS) unit. They will apply the the patches of the TENS unit around the C-section site. Starting 8 hours after C-Section, the TENS unit will be turned on and will remain on until the patient is discharged, to be removed for toilet and showering at the patient's discretion. Once the TENS unit is applied and turned on, the patient will not have to do anything else to maintain the therapy. Routine pharmacologic care will also be available.
  Interventions: Device: Transcutaneous Electrical Nerve Stimulation (TENS)
- Opioid Addicted Post-CS TENS (Experimental): Subjects will be targeted on the basis of opioid addiction and usage of methadone maintenance. The patients in the intervention group will be educated on the proper way to utilize the transcutaneous electrical nerve stimulation (TENS) unit. They will apply the the patches of the TENS unit around the C-section site). Starting 8 hours after C-Section, the TENS unit will be turned on and will remain on until the patient is discharged, to be removed for toilet and showering at the patient's discretion. Once the TENS unit is applied and turned on, the patient will not have to do anything else to maintain the therapy. Routine pharmacologic care will also be available.
  Interventions: Device: Transcutaneous Electrical Nerve Stimulation (TENS)
- Post-CS Routine Care (No Intervention): Routine pharmacologic care will be provided.
- Opioid Addicted Post-CS Routine Care (No Intervention): Routine pharmacologic care will be provided.

INTERVENTIONS:
Device: Transcutaneous Electrical Nerve Stimulation (TENS) — Starting 8 hours after cesarean section, the TENS unit will be applied with charges above and below the incision. The device will be set to high frequency (>75 Hz) for pain relief. Intensity of stimulation will be set to patient threshold using the forearm as a guide. Stimulation will be turned on titrated to the level which is felt but not painful for the patient. It will remain on until the patient is discharged, to be removed for toilet and showering at the patient's discretion. Once the TENS unit is applied and turned on, the patient will not have to do anything else to maintain the therapy.
  Arms: Opioid Addicted Post-CS TENS; Post-CS TENS

SUMMARY:
We propose to explore the effects of Transcutaneous Electrical Nerve Stimulation (TENS) therapy in the pain management of postpartum women.

A. Objectives

* To determine if the addition of TENS therapy to the pain management of women post-cesarean section leads to less opioid medication use.
* To evaluate the efficacy of TENS therapy as a means of alternative pain relief for women post-cesarean section with a history of opioid use.

B. Hypotheses / Research Question(s) We hypothesize that patients that receive TENS therapy will report lower pain scores and request less opioid medication than the control group. We anticipate improved control in particular in the group of women with a history of opioid use.

Additionally, we believe that the TENS therapy will show benefits in other postpartum outcomes including time to bowel movement, level of sedation, and time to out of bed.

Overall, we anticipate that this pilot study will support the application of TENS therapy in postpartum pain management.

DETAILED DESCRIPTION:
OVERVIEW. This study is a pilot randomized interventional trial. Two categories of participants will be randomly assigned to an invention or control group, using a random number generator: normal cesarean without associated comorbidity, or cesarean in women with a history of opioid addiction. The control group will receive usual care. The intervention group will receive usual care plus TENS therapy beginning 8 hours after cesarean section and continuing to discharge. Both groups will receive medications for pain as requested or ordered by the doctor.

RESEARCH PROCEDURES. Patients will be identified for participation in their prenatal visit, and will be approached for study inclusion. Physicians that have a direct treatment relationship with the patient will inform the patient about the study and invite them to enroll. Consent for participation will be reviewed with the principal investigator and signed prior to delivery hospitalization. Randomization will follow consent, and patients randomized to intervention will have teaching performed about how to use the device at the time of consent.

Following cesarean delivery, subjects will be re-approached in the Postpartum Unit at Robert Wood Johnson University Hospital by study staff. The TENS device will be again reviewed, and provided to the patient, with review of instructions for use. The patients in the intervention group will be educated on the proper way to utilize the TENS unit. They will apply the the patches of the TENS unit around the C-section site. Starting 8 hours after C-Section, the TENS unit will be turned on and will remain on until the patient is discharged, to be removed for toilet and showering at the patient's discretion. Once the TENS unit is applied and turned on, the patient will not have to do anything else to maintain the therapy. Study staff will provide a record for documentation of time on/off for the unit. On the day of discharge, study staff will collect the device, and conduct a short survey about pain score. They will then review pain scores, pain medication usage and other secondary outcomes in the patient's chart. Finally, pain will be reassessed at the subject's outpatient postpartum visits by study staff.

DATA COLLECTION. Our research team members will collect the following data points from the patient's inpatient medical record: pain scale scores, medication requests/prescriptions (including name, type, and amount), time to first bowel movement, subjective incision complaints, and time to OOB. Participants will complete a survey before discharge which will solicit additional information about the postpartum recovery experience with or without TENS therapy.

DURATION OF STUDY. Study duration will be no more than 12 weeks. This will include up to 6 weeks prior to delivery for study approach and consent, delivery hospitalization, and 6 weeks postpartum for pain assessments at postpartum visits. There will be no long term follow up.

PRIMARY and SECONDARY ENDPOINTS. Primary endpoint of this pilot study is a total of 10 normal patients undergoing cesarean, and 10 patients with history of opioid addiction. Intervention will be performed in 5 patients in each group. Safety data will be reviewed following the first 10 patients to evaluate for worsening patient scores relative to controls.

ELIGIBILITY:
Inclusion Criteria:

* Women aged between 18 and 45 years
* Understand and be able to follow written and oral instructions in English
* Provide written informed consent
* History of prior opioid addiction for half of the patients.

Exclusion Criteria:

- History of cardiac arrhythmia or pacemaker usage

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2018-11-09 (Actual); Primary Completion 2020-01-31 (Actual); Study Completion 2020-03-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Adrienne Simonds, PT PhD, Principal Investigator — Rutgers School of Health Professions
Locations (1):
- Robert Wood Johnson University Hospital, New Brunswick, New Jersey, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Dowell D, Haegerich TM, Chou R. CDC Guideline for Prescribing Opioids for Chronic Pain--United States, 2016. JAMA. 2016 Apr 19;315(15):1624-45. doi: 10.1001/jama.2016.1464. PMID 26977696
- [Background] Hollinger JL. Transcutaneous electrical nerve stimulation after cesarean birth. Phys Ther. 1986 Jan;66(1):36-8. doi: 10.1093/ptj/66.1.36. PMID 3484553
- [Background] Citak Karakaya I, Yuksel I, Akbayrak T, Demirturk F, Karakaya MG, Ozyuncu O, Beksac S. Effects of physiotherapy on pain and functional activities after cesarean delivery. Arch Gynecol Obstet. 2012 Mar;285(3):621-7. doi: 10.1007/s00404-011-2037-0. Epub 2011 Aug 10. PMID 21830007
- [Background] Kayman-Kose S, Arioz DT, Toktas H, Koken G, Kanat-Pektas M, Kose M, Yilmazer M. Transcutaneous electrical nerve stimulation (TENS) for pain control after vaginal delivery and cesarean section. J Matern Fetal Neonatal Med. 2014 Oct;27(15):1572-5. doi: 10.3109/14767058.2013.870549. Epub 2014 Jan 8. PMID 24283391
- [Background] Osmundson SS, Schornack LA, Grasch JL, Zuckerwise LC, Young JL, Richardson MG. Postdischarge Opioid Use After Cesarean Delivery. Obstet Gynecol. 2017 Jul;130(1):36-41. doi: 10.1097/AOG.0000000000002095. PMID 28594766
- [Background] Reynolds RA, Gladstone N, Ansari AH. Transcutaneous electrical nerve stimulation for reducing narcotic use after cesarean section. J Reprod Med. 1987 Nov;32(11):843-6. PMID 2892930
- [Background] Smith CM, Guralnick MS, Gelfand MM, Jeans ME. The effects of transcutaneous electrical nerve stimulation on post-cesarean pain. Pain. 1986 Nov;27(2):181-193. doi: 10.1016/0304-3959(86)90209-5. PMID 3540813
- [Background] Willmann S, Edginton AN, Coboeken K, Ahr G, Lippert J. Risk to the breast-fed neonate from codeine treatment to the mother: a quantitative mechanistic modeling study. Clin Pharmacol Ther. 2009 Dec;86(6):634-43. doi: 10.1038/clpt.2009.151. Epub 2009 Aug 26. PMID 19710640

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Post-CS TENS | Opioid Addicted Post-CS TENS | Post-CS Routine Care | Opioid Addicted Post-CS Routine Care
Started | 5 | 3 | 5 | 2
Completed | 5 | 3 | 5 | 2
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Post-CS TENS | Opioid Addicted Post-CS TENS | Post-CS Routine Care | Opioid Addicted Post-CS Routine Care | Total
Number analyzed (Participants) | 5 | 3 | 5 | 2 | 15
Age, Categorical [Count of Participants; unit: Participants] — Participants were between 18 and 45 years to be eligible. Participant age was not retained after determining eligibility for enrollment.
  Participants
    <=18 years | 0 | 0 | 0 | 0 | 0
    Between 18 and 65 years | 5 | 3 | 5 | 2 | 15
    >=65 years | 0 | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants] — All participants were female. Males were excluded from this study.
  Participants
    Female | 5 | 3 | 5 | 2 | 15
    Male | 0 | 0 | 0 | 0 | 0
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants] — All participants received prenatal care from the Rutgers Medical Group Obstetrics and Gynecology or Maternal Fetal Medicine practices and the High Risk Obstetric Perinatal Clinic and delivered via Cesarean Section at Robert Wood Johnson University Hospital in New Brunswick, New Jersey, United States.
  participants
    United States | 5 | 3 | 5 | 2 | 15
History of prior opioid addiction [Count of Participants; unit: Participants] — A history of opioid addiction was sought for half the patients in this trial.
  Participants | 0 | 3 | 0 | 2 | 5
Cesarean section delivery [Count of Participants; unit: Participants] — All participants delivered via Cesarean Section.
  Participants | 5 | 3 | 5 | 2 | 15

OUTCOME MEASURES:

1. Primary Outcome: Post-operative Pain Ratings
Description: Post-operative pain rating (0-10 scale) using Visual Analog Scale (VAS). VAS scores correspond self-report pain intensity. Higher scores mean higher pain intensity.
Time Frame: 3-4 post-operative days
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Post-CS TENS | Opioid Addicted Post-CS TENS | Post-CS Routine Care | Opioid Addicted Post-CS Routine Care
Number analyzed (Participants) | 5 | 3 | 5 | 2
units on a scale | 2.90 (1.9) | 3.7 (2.97) | 2.58 (2.29) | 4.24 (2.9)

2. Secondary Outcome: Milligrams Morphine Equivalent
Description: Milligrams morphine equivalent (MME) is a standardized method of totaling dose of opioid medication. MME uses a conversion factor to convert opioid medication dosages into morphine equivalents, in milligrams.
Time Frame: 3-4 post-operative days
Measure: Mean (Standard Deviation); unit: Milligrams
Arm/Group | Post-CS TENS | Opioid Addicted Post-CS TENS | Post-CS Routine Care | Opioid Addicted Post-CS Routine Care
Number analyzed (Participants) | 5 | 3 | 5 | 2
Milligrams | 58.5 (18.67) | 182.83 (112.79) | 57 (35.42) | 105 (84.85)

3. Secondary Outcome: Acetominophen Dosage
Description: Total dosage of acetominophen in milligrams. Acetominophen is a non-opioid analgesic medication.
Time Frame: 3-4 postoperative days
Measure: Mean (Standard Deviation); unit: Milligrams
Arm/Group | Post-CS TENS | Opioid Addicted Post-CS TENS | Post-CS Routine Care | Opioid Addicted Post-CS Routine Care
Number analyzed (Participants) | 5 | 3 | 5 | 2
Milligrams | 3335 (578.68) | 3750 (3031.08) | 1955 (1502.96) | 5050 (4384.06)

4. Secondary Outcome: Ibuprofen Dosage
Description: Total ibuprofen dosage in milligrams. Ibuprofen is a non-steroidal anti-inflammatory (NSAID) medication used to reduce pain and inflammation.
Time Frame: 3-4 postoperative days
Measure: Mean (Standard Deviation); unit: Milligrams
Arm/Group | Post-CS TENS | Opioid Addicted Post-CS TENS | Post-CS Routine Care | Opioid Addicted Post-CS Routine Care
Number analyzed (Participants) | 5 | 3 | 5 | 2
Milligrams | 4680 (1154.12) | 1400 (916.52) | 4500 (774.6) | 4500 (1272.79)

5. Secondary Outcome: Time to OOB
Description: Time to get out of bed (OOB) measured in hours
Time Frame: 3-4 post-operative days
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Post-CS TENS | Opioid Addicted Post-CS TENS | Post-CS Routine Care | Opioid Addicted Post-CS Routine Care
Number analyzed (Participants) | 5 | 3 | 5 | 2
hours | 11.2 (6.3) | 16.7 (2.1) | 14.4 (6.5) | 20.0 (1.4)

6. Secondary Outcome: Time to First BM
Description: Time to first bowel movement (BM) measured in hours
Time Frame: 3-4 post-operative days
Population: This data were not collected due to unanticipated error.
Arm/Group | Post-CS TENS | Opioid Addicted Post-CS TENS | Post-CS Routine Care | Opioid Addicted Post-CS Routine Care
Number analyzed (Participants) | 0 | 0 | 0 | 0

7. Secondary Outcome: Level of Sedation
Description: Level of sedation (0-10 scale) was measured by provider observation via a Visual Analogue Scale. Higher scores mean more sedation.
Time Frame: 3-4 post-operative days
Population: This data were not collected due to unanticipated error.
Arm/Group | Post-CS TENS | Opioid Addicted Post-CS TENS | Post-CS Routine Care | Opioid Addicted Post-CS Routine Care
Number analyzed (Participants) | 0 | 0 | 0 | 0

8. Secondary Outcome: Number of Participants Who Found the Device Acceptable
Description: Device acceptability questionnaire asked participants in the intervention group if TENS positively impacted their recovery. Responses indicated the number of participants who indicated "Yes" that TENS positively impacted their recovery. Responses of "Unsure" or "No" were coded as "No" responses.
Time Frame: 3-4 days postoperatively
Measure: Count of Participants; unit: Participants
Arm/Group | Post-CS TENS | Opioid Addicted Post-CS TENS | Post-CS Routine Care | Opioid Addicted Post-CS Routine Care
Number analyzed (Participants) | 5 | 2 | 5 | 2
Participants | 3 | 1 | 0 | 0

9. Secondary Outcome: McGill Pain Questionnaire
Description: The Short-Form McGill Pain Questionnaire (SFMPQ) includes 15 items that describe the type of pain from sensory and affective domains. Each item is scored 0 to 3, with scores>1 indicating that pain aligns with that descriptor. Higher scores indicate more severe symptoms. The score range is 0 to 78, with 78 representing more severe pain.
Time Frame: 3-4 days postoperatively
Measure: Mean (Full Range); unit: score on a scale
Arm/Group | Post-CS TENS | Opioid Addicted Post-CS TENS | Post-CS Routine Care | Opioid Addicted Post-CS Routine Care
Number analyzed (Participants) | 5 | 2 | 4 | 2
score on a scale | 7.8 [3 to 13] | 19 [11 to 27] | 10 [4 to 14] | 19 [18 to 20]

10. Secondary Outcome: Neuropathic Pain Scale (NPS)
Description: Neuropathic Pain Scale (NPS) is a 10-item self-questionnaire that measures the degree of neuropathic pain. Higher scores indicate more severe pain. Total score ranges from 0 to 100, with 100 indicating the most severe neuropathic pain. Total NPS score is reported.
Time Frame: 3-4 postoperative days
Measure: Mean (Full Range); unit: score on a scale
Arm/Group | Post-CS TENS | Opioid Addicted Post-CS TENS | Post-CS Routine Care | Opioid Addicted Post-CS Routine Care
Number analyzed (Participants) | 4 | 3 | 4 | 2
score on a scale | 22.4 [9 to 35] | 49 [49 to 49] | 24.875 [8 to 32.5] | 64.5 [58 to 71]

11. Secondary Outcome: Acceptability Questionnaire
Description: Device acceptability questionnaire included 5 total self-report questions. Device usage (time used) and discharge medications were text entry questions. Three yes/no questions asked about impacts on pain relief, recovery and breastfeeding.
Time Frame: 6 weeks postoperatively
Population: Data was not collected because participants could not be reached.
Arm/Group | Post-CS TENS | Opioid Addicted Post-CS TENS | Post-CS Routine Care | Opioid Addicted Post-CS Routine Care
Number analyzed (Participants) | 0 | 0 | 0 | 0

12. Secondary Outcome: McGill Pain Questionnaire
Description: The Short-Form McGill Pain Questionnaire (SFMPQ) includes 15 items that describe the type of pain from sensory and affective domains. Each item is scored 0 to 3, with scores>1 indicating that pain aligns with that descriptor. Higher scores indicate more severe symptoms.
Time Frame: 6 weeks postoperatively
Population: Data was not collected because participants could not be reached.
Arm/Group | Post-CS TENS | Opioid Addicted Post-CS TENS | Post-CS Routine Care | Opioid Addicted Post-CS Routine Care
Number analyzed (Participants) | 0 | 0 | 0 | 0

13. Secondary Outcome: Neuropathic Pain Scale
Description: Neuropathic Pain Scale (NPS) is a 10-item questionnaire that measures the degree of neuropathic pain. Higher scores indicate more severe pain.
Time Frame: 6 weeks postoperatively
Population: Data was not collected because participants could not be reached.
Arm/Group | Post-CS TENS | Opioid Addicted Post-CS TENS | Post-CS Routine Care | Opioid Addicted Post-CS Routine Care
Number analyzed (Participants) | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Adverse event data were collected for the duration of the postpartum inpatient hospital stay, generally 3 to 4 days.
Description: There were no adverse events reported.
Arm/Group | Post-CS TENS | Opioid Addicted Post-CS TENS | Post-CS Routine Care | Opioid Addicted Post-CS Routine Care
All-Cause Mortality (participants affected / at risk) | 0/5 | 0/3 | 0/5 | 0/2
Serious Adverse Events (participants affected / at risk) | 0/5 | 0/3 | 0/5 | 0/2
Other Adverse Events (participants affected / at risk) | 0/5 | 0/3 | 0/5 | 0/2

LIMITATIONS AND CAVEATS:
Early termination of study because of COVID-19 pandemic limited number of enrolled subjects.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol (2022-07-19): https://cdn.clinicaltrials.gov/large-docs/88/NCT03843788/Prot_002.pdf
  • Statistical Analysis Plan (2024-07-11): https://cdn.clinicaltrials.gov/large-docs/88/NCT03843788/SAP_005.pdf
  • Informed Consent Form (2020-08-26): https://cdn.clinicaltrials.gov/large-docs/88/NCT03843788/ICF_004.pdf